CLINICAL TRIAL: NCT00492765
Title: A Multi-centre, Double Blind, Randomised, Placebo Controlled, Parallel Group Study Investigating Simvastatin as an Add-on Treatment IM Administered Interferon-beta-1a for the Treatment of Relapsing-Remitting Multiple Sclerosis
Brief Title: Simvastatin as an Add-on Treatment to Interferon-beta-1a for the Treatment of Relapsing-Remitting Multiple Sclerosis
Acronym: SIMCOMBIN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Biogen Idec MD, Biogen Idec
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SIMCOMBIN
Record Dates: First submitted 2007-06-25; First posted 2007-06-27 (Estimated); Last update posted 2010-10-15 (Estimated); Status verified 2010-10

CONDITIONS: Multiple Sclerosis
Keywords: Combination therapy; Simvastatin; Multiple Sclerosis; Interferon-beta-1a
MeSH Terms: conditions — Multiple Sclerosis | interventions — Interferon beta-1a; Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): interferon beta-1a and Simvastatin
  Interventions: Drug: Interferon-beta-1a; Drug: Simvastatin
- 2 (Placebo Comparator): Interferon beta-1a and Placebo
  Interventions: Drug: Interferon-beta-1a; Drug: Placebo

INTERVENTIONS:
Drug: Interferon-beta-1a — dosage and frequency as per label
  Other Names: Avonex
Drug: Simvastatin — dosage and frequency as per Biogen Idec protocol
  Arms: 1
Drug: Placebo — dosage and frequency the same as simvastatin as per Biogen Idec Protocol
  Arms: 2

SUMMARY:
This study is to find out if there is any benefit to adding Simvastatin to Interferon-beta-1a in patients with Multiple Sclerosis.

DETAILED DESCRIPTION:
This is a multi-centre, double blind, placebo controlled, randomised, parallel group, phase 4 study. Following three months treatment with Interferon beta 1a (Avonex) patients will be randomised for treatment with simvastatin or placebo as an add-on to interferon -beta-1a (AvonexÒ). Patients will start treatment with 40 mg peroral simvastatin daily or identically appearing placebo for one month. Hereafter, patients will escalate dosage to 80 mg daily. The patients will be examined clinically at baseline and at, 3, 4, 6, 9, 12 and 15 months. Patients who attend visit 5 (15 months) before the last patient has attended this visit will be asked to attend additional visits (visits 6+) until the last patient has attended visit 5. Clinical examination will be performed, for applicable patients, at 3 month intervals until the end of the study. This will be a maximum of two years, i.e. no more than eight additional visits. Laboratory assessments will be performed at screening 3, 4, 6, 9, 12 and 15 months after baseline, and for applicable patients additionally at 3 month intervals until end of study. MRI will be performed (T1-weighted and T2-weighted) at randomisation (3 months after baseline) and 12 months hereafter.

ELIGIBILITY:
Inclusion Criteria:

* Is between the age of 18 and 55 years (both included)
* Relapsing-remitting MS according to Poser criteria (CDMS or LSDMS) 22 or definite MS according to McDonald criteria 23
* Disability equivalent to an EDSS of 5.5 or less 21
* Clinical activity defined as at least one reported or documented relapse within the last year
* Patient must be prepared to and considered able to follow the protocol during the whole study period and to attend the planned visits, even if the treatment has to be withdrawn

Exclusion Criteria:

* Any condition that might give rise to similar symptoms as MS
* Immunomodulatory or immunosuppressive treatment for MS prior to inclusion into the study (prior pulse steroid treatment for relapses is allowed)
* Treatment with glucocorticoids or ACTH later than one month prior to inclusion into the study, i.e. at the screening visit
* Onset of a relapse within one month prior to inclusion into the study, i.e. at the screening visit
* History of major depression
* Alcohol or drug dependency
* Cardiac insufficiency, cardiomyopathy, significant cardiac dysrhythmia, unstable or advanced ischemic heart disease (NYHA III or IV)
* Significant hypertension (BP > 180/110 mmHg)
* Renal insufficiency defined as serum creatinine > 1.5 times the upper normal reference limit
* Total plasma cholesterol < 3.5 mmol/L
* Any medical illness requiring treatment with systemic corticosteroids
* Any systemic disease that can influence the patient's safety and compliance, or the evaluation of the disability
* Women who are pregnant, breast-feeding or have the possibility for pregnancy during the study. To avoid pregnancy, women have to be postmenopausal, surgically sterile, sexually inactive or practice reliable contraception

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 380 (Actual)
Dates: Start 2006-02; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
The time to first documented relapse | months 4, 6, 9, 12, and every 3 months from months 18-39

SECONDARY OUTCOMES:
3Annual rate of documented relapses after randomisation | months 4, 6, 9, 12, and every 3 months from months 18-39
Number of new and/or enlarging lesions on T2-weighted MRI based on MRI done 12 months following randomisation compared with MRI done at time of randomisation | month 15
Proportion of patients without disease activity after randomisation (i.e. no relapses, no increase in EDSS score and no increase in enlarging or new T2 lesions). | months 4, 6, 9, 12, and every 6 months from months 18-39

CONTACTS AND LOCATIONS:
Locations (1):
- Coordinating Research Site, Copenhagen, Denmark

REFERENCES:
- [Derived] Sorensen PS, Lycke J, Eralinna JP, Edland A, Wu X, Frederiksen JL, Oturai A, Malmestrom C, Stenager E, Sellebjerg F, Sondergaard HB; SIMCOMBIN study investigators. Simvastatin as add-on therapy to interferon beta-1a for relapsing-remitting multiple sclerosis (SIMCOMBIN study): a placebo-controlled randomised phase 4 trial. Lancet Neurol. 2011 Aug;10(8):691-701. doi: 10.1016/S1474-4422(11)70144-2. PMID 21742556